CLINICAL TRIAL: NCT03356262
Title: The QUebec Adipose and Lifestyle InvesTigation in Youth (QUALITY) Cohort
Acronym: QUALITY
Status: Active, not recruiting | Type: Observational
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Melanie Henderson, Clinical assistant professor, St. Justine's Hospital
Other Study IDs: QUALITY
Record Dates: First submitted 2017-11-11; First posted 2017-11-29 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Obesity, Childhood; Diabetes Mellitus, Type 2; Cardiovascular Risk Factor; Pediatric ALL; Lifestyle; Physical Activity; Sedentary Lifestyle; Diet Habit; Metabolic Complication
Keywords: Cohort study
MeSH Terms: conditions — Pediatric Obesity; Diabetes Mellitus, Type 2; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Motor Activity; Sedentary Behavior; Feeding Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, blood, serum, urine, stool, saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The QUebec Adipose and Lifestyle InvesTigation in Youth (QUALITY) Cohort study is a unique and comprehensive longitudinal study of 630 Caucasian children and their parents that was designed to investigate the natural history and determinants of childhood obesity and its cardiometabolic consequences.

DETAILED DESCRIPTION:
The QUALITY Cohort is funded by the Canadian Institutes of Health Research, the Heart and Stroke Foundation of Canada, as well as the Fonds de la recherche en santé du Québec. The multidisciplinary study team comprises over 20 researchers with a wide variety of relevant expertise as well as research fellows, students and staff (www.etudequalitystudy.ca).

The specific objectives of QUALITY are: 1) To increase understanding of the natural history of excess weight and its associated cardiometabolic consequences (dyslipidemia, hyperinsulinemia, dysglycemia, inflammation, elevated blood pressure, sympathetic overactivity) in youth at risk for the development of obesity; 2) To investigate the relative importance of the genetic, biological, environmental and psychosocial determinants of excess weight and its associated cardiometabolic consequences. Determinants of particular interest include social factors (socio-economic status, family composition, built environment), behavioural factors (eating behaviour, physical activity, smoking, sleep, stress), biological factors (adverse fetal environment, body fat distribution, growth trajectory, aerobic fitness), metabolic factors (insulin sensitivity, adipocytokines), and genetic/familial factors (family history, parental characteristics, gene variations); 3) To examine the relation between obesity, cardiometabolic complications, and subclinical markers of atherosclerosis; and 4) To examine whether obesity and its associated risk factor are related to children's oral health.

The QUALITY Cohort used a school-based sampling strategy to identify potential participants. About 400 000 recruitment flyers were distributed over three consecutive years to parents of children in Grades 2 to 5, in 1040 primary schools (89% of schools approached) including 44 private schools situated within 75 km of Montreal, Quebec City and Sherbrooke in the province of Quebec, Canada. Families interested in participating were invited to contact the research coordinator for additional information, to confirm eligibility, and to set an appointment with the research team; 1320 of 3350 families who contacted the coordinator met the inclusion criteria. Six hundred and thirty families agreed to participate and completed the baseline evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 8-10 years at baseline;
* Caucasian of Western European ancestry;
* At least one obese biological parent (i.e., body mass index (BMI) ≥30 kg/m2 or waist circumference >102 cm in men and >88 cm in women, based on self-reported measurements of height, weight and waist circumference)
* Both biological parents available to participate in the baseline assessment.

Exclusion Criteria:

* Children with a previous diagnosis of Type 1 or 2 diabetes;
* Children with a previous diagnosis of a serious illness, psychological condition, or cognitive disorder which hindered participation in some or all of the study components;
* Children treated with anti-hypertensive medication or steroids (except if administered topically or through inhalation);
* Children following a very restricted diet (< 600 kcal/day);
* Mother pregnant or breastfeeding at the baseline evaluation;
* Family with pending plans to move out of the province of Quebec (Canada).

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 630 Caucasian families with a child aged 8-10 years agreed to participate and completed the baseline evaluation.
  564 families completed the second round of data collection 2 years later. 377 families completed the third round of data collection 7 years after the baseline assessment.
  A 4th round of data collection is currently being prepared.
Sampling Method: Non-Probability Sample
Enrollment: 630 (Actual)
Dates: Start 2005-07-25 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Body mass index (BMI) | Through study completion, 13 - 14 years post baseline
  Weight (kg) and height (m) will be combined to report BMI in kg/m^2 and transformed to z-scores using WHO standards

SECONDARY OUTCOMES:
Waist circumference | Through study completion, 13 - 14 years post baseline
  Measured in centimeters, midway between the last floating rib and the iliac crest
% body fat mass | Through study completion, 13 - 14 years post baseline
  Measured using dual energy x-ray absorptiometry and combined as total body fat mass in kg / total body mass in kg * 100
Impaired fasting glucose | Through study completion, 13 - 14 years post baseline
  Measured from a blood sample collected using venipuncture following a 12-hour overnight fast. Plasma glucose concentrations were computed on the Beckman Coulter Synchron LX20 automat using the glucose oxidase method. Analyses were performed in batches at the Centre Hospitalier Universitaire Sainte-Justine Clinical Biochemistry laboratory twice monthly. Considered as impaired fasting blood glucose if greater or equal to 5.6 mmol/L.
Impaired glucose tolerance | Through study completion, 13 - 14 years post baseline
  Participants underwent a 2-hour oral glucose tolerance test (OGTT) after a 12-hour overnight fast. Blood samples were collected at 30-, 60-, 90-, and 120-minute intervals after an oral glucose dose of 1.75 g/kg of body weight (maximum 75 g). Plasma glucose concentrations were computed on the Beckman Coulter Synchron LX20 automat using the glucose oxidase method. Analyses were performed in batches at the Centre Hospitalier Universitaire Sainte-Justine Clinical Biochemistry laboratory twice monthly. Considered as impaired glucose tolerence blood glucose at 2hrs of the OGTT greater or equal to 7.8 mmol/L.
Type 2 diabetes | Through study completion, 13 - 14 years post baseline
  Type 2 diabetes was diagnosed according to recognized criteria from the Canadian Diabetes Association (Canadian Diabetes Association Clinical Practice Guidelines Expert Committee. Canadian Diabetes Association 2013 Clinical Practice Guidelines for the Prevention and Management of Diabetes in Canada. Can J Diabetes 2013;37(suppl 1):S1-S212.)
Hypertension (systolic) | Through study completion, 13 - 14 years post baseline
  Systolic and diastolic blood pressures (SBP and DBP, respectively) were measured using an appropriately sized arm cuff and an automated oscillometric blood pressure monitor doing 5 repeat measures at 1 min intervals (Dinamap model CR9340). Participants were seated and had to rest for 5 minutes prior to the measurement. The average of the last three measures of SBP and DBP was used in the analyses. These were then transformed to age-, sex-, and height-specific Z-scores according to The Fourth Report on the Diagnosis, Evaluation, and Treatment of High Blood Pressure in Children and Adolescents. Considered hypertensive if SBP > 95th percentile for age, sex, and height.
Hypertension (diastolic) | Through study completion, 13 - 14 years post baseline
  Systolic and diastolic blood pressures (SBP and DBP, respectively) were measured using an appropriately sized arm cuff and an automated oscillometric blood pressure monitor doing 5 repeat measures at 1 min intervals (Dinamap model CR9340). Participants were seated and had to rest for 5 minutes prior to the measurement. The average of the last three measures of SBP and DBP was used in the analyses. These were then transformed to age-, sex-, and height-specific Z-scores according to The Fourth Report on the Diagnosis, Evaluation, and Treatment of High Blood Pressure in Children and Adolescents. Considered hypertensive if DBP > 95th percentile for age, sex, and height.
Dyslipidemia | Through study completion, 13 - 14 years post baseline
  Blood samples were obtained by venipuncture after a 12 hour overnight fast. Lipids (high density lipoprotein (HDL) cholesterol and triglycerides) were measured on a Synchron LX®20 analyzer, with Beckman Instruments reagents, by the Department of Clinical Biochemistry at CHU Sainte-Justine, according to the recommendations of the International Federation of Clinical Chemistry. Low density lipoprotein (LDL) cholesterol was calculated based on the Friedewald equation. Dyslipedimia was defided according to published guidelines (Pediatrics. 2011 Dec; 128(Suppl 5): S213-S256.)

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Henderson, MD, PhD, Principal Investigator — Université de Montréal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lambert M, Van Hulst A, O'Loughlin J, Tremblay A, Barnett TA, Charron H, Drapeau V, Dubois J, Gray-Donald K, Henderson M, Lagace G, Low NC, Mark S, Mathieu ME, Maximova K, McGrath JJ, Nicolau B, Pelletier C, Poirier P, Sabiston C, Paradis G. Cohort profile: the Quebec adipose and lifestyle investigation in youth cohort. Int J Epidemiol. 2012 Dec;41(6):1533-44. doi: 10.1093/ije/dyr111. Epub 2011 Jul 23. No abstract available. PMID 21785124
- [Derived] Saade MB, Holden S, Kakinami L, McGrath JJ, Mathieu ME, Poirier P, Barnett TA, Beaucage P, Henderson M. Adiposity and cardiac autonomic function in children with a family history of obesity. Clin Auton Res. 2024 Dec;34(6):583-592. doi: 10.1007/s10286-024-01063-y. Epub 2024 Sep 21. PMID 39304555
- [Derived] Harnois-Leblanc S, Van Hulst A, Lucibello KM, Harbec MJ, Sabiston CM, Maximova K, Sylvestre MP, Henderson M. Associations Between Weight-Loss Attempts, Weight-Related Stress, and Body Image During Childhood and Adolescence in Children With Parental Obesity. Child Obes. 2024 Sep;20(6):434-441. doi: 10.1089/chi.2023.0082. Epub 2024 Jan 19. PMID 38241489
- [Derived] Sohi DK, Van Hulst A, McNealis V, Simoneau G, Drapeau V, Barnett TA, Mathieu ME, Paradis G, Tremblay A, Benedetti A, Henderson M. Early Lifestyle Determinants of Adiposity Trajectories from Childhood into Late Adolescence. Child Obes. 2024 Jul;20(5):336-345. doi: 10.1089/chi.2023.0062. Epub 2023 Dec 13. PMID 38100098
- [Derived] Roberge JB, Harnois-Leblanc S, McNealis V, van Hulst A, Barnett TA, Kakinami L, Paradis G, Henderson M. Body Mass Index Z Score vs Weight-for-Length Z Score in Infancy and Cardiometabolic Outcomes at Age 8-10 Years. J Pediatr. 2021 Nov;238:208-214.e2. doi: 10.1016/j.jpeds.2021.07.046. Epub 2021 Jul 21. PMID 34302856
- [Derived] Van Hulst A, Paradis G, Harnois-Leblanc S, Benedetti A, Drapeau V, Henderson M. Lowering Saturated Fat and Increasing Vegetable and Fruit Intake May Increase Insulin Sensitivity 2 Years Later in Children with a Family History of Obesity. J Nutr. 2018 Nov 1;148(11):1838-1844. doi: 10.1093/jn/nxy189. PMID 30383280
- [Derived] Roberge JB, Van Hulst A, Barnett TA, Drapeau V, Benedetti A, Tremblay A, Henderson M. Lifestyle Habits, Dietary Factors, and the Metabolically Unhealthy Obese Phenotype in Youth. J Pediatr. 2019 Jan;204:46-52.e1. doi: 10.1016/j.jpeds.2018.08.063. Epub 2018 Oct 23. PMID 30366774
- [Derived] Van Hulst A, Paradis G, Benedetti A, Barnett TA, Henderson M. Pathways Linking Birth Weight and Insulin Sensitivity in Early Adolescence: A Double Mediation Analysis. J Clin Endocrinol Metab. 2018 Dec 1;103(12):4524-4532. doi: 10.1210/jc.2018-00525. PMID 30137396